CLINICAL TRIAL: NCT07144956
Title: Is Adding Cilostazol to Nimodipine Improving Neurological Outcome of Patients With Aneurysmal Subarachnoid Hemorrhage? A Randomized, Double Blind, Placebo-controlled Trial
Brief Title: Cilostazol With Nimodipine to Improve Outcome After Aneurysmal Subarachnoid Hemorrhage
Acronym: CASH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D24-009; 2024-516468-27-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-04; First posted 2025-08-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Cilostazol; Nimodipine; Vasospasm; Modified Rankin Scale (mRS); Neurological outcome; Double-blind; Randomized Controlled Trial; Multicenter clinical trial
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Cilostazol

STUDY DESIGN:
Intervention Model Description: The CASH study is a phase III, multicenter, randomized, double-blind, placebo-controlled clinical trial with a parallel-group, adaptive sequential design. Adult patients admitted to intensive care within 96 hours of an aneurysmal subarachnoid hemorrhage (aSAH), and after successful aneurysm securing (clipping or coiling), are randomized into two groups. The experimental group receives cilostazol (100 mg twice daily for 14 days) in addition to standard nimodipine (21 days), while the control group receives placebo plus nimodipine. The primary objective is to assess neurological outcome at 6 months using the modified Rankin Scale. The total study duration is 49 months, including 42 months of enrollment and 6 months of follow-up. Two interim analyses are planned. The study is funded by a PHRC and monitored by an independent Data Safety Monitoring Board (DSMB).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cilostazol + Nimodipine (Experimental): In the cilostazol arm, patients will receive standard care for aneurysmal subarachnoid hemorrhage, including nimodipine administration as recommended by French and European guidelines for delayed cerebral ischemia (DCI) prevention. In addition, participants will receive cilostazol 100 mg twice daily, administered orally or via gastric tube if swallowing is not possible, for 14 consecutive days, starting within 96 hours of hemorrhage onset. Cilostazol tablets may be crushed for enteral administration. All other preventive and curative treatments for vasospasm or DCI-such as hypertensive therapy, milrinone, or endovascular interventions-are permitted at the discretion of the treating physician. Monitoring will include clinical status, occurrence of vasospasm, DCI, cerebral infarction, and cilostazol-related adverse events. Follow-up visits and safety assessments will be identical to the placebo arm.
  Interventions: Biological: Cilostazol (Pletal®) 100 mg Tablets; Drug: Nimodipine group
- Nimodipine + Placebo (Placebo Comparator): In the placebo arm, patients will receive standard care for aneurysmal subarachnoid hemorrhage, which must include nimodipine for the prevention of delayed cerebral ischemia (DCI) as per French and European guidelines. Nimodipine will be administered orally/enterally or intravenously, with dose, route, and duration decided by the treating physician according to patient status and local practice. Participants will receive a placebo, visually identical to cilostazol tablets, given orally or via gastric tube twice daily for 14 days, starting within 96 hours of hemorrhage onset. All other preventive or curative treatments for vasospasm or DCI-such as hypertensive therapy, milrinone, or endovascular procedures-are allowed at the physician's discretion. Monitoring, follow-up, and safety assessments will be performed in the same manner as in the experimental arm.
  Interventions: Drug: Placebo; Drug: Nimodipine group

INTERVENTIONS:
Biological: Cilostazol (Pletal®) 100 mg Tablets — 100 mg orally or via feeding tube twice daily for 14 days, starting within 96 hours after aneurysmal subarachnoid hemorrhage onset. Tablets may be crushed for enteral administration.
  Arms: Cilostazol + Nimodipine
Drug: Placebo — Oral or enteral placebo, visually identical to cilostazol, twice daily for 14 days, starting within 96 hours after hemorrhage onset.
  Other Names: Placebo (matching Cilostazol)
  Arms: Nimodipine + Placebo
Drug: Nimodipine group — Administered orally, enterally, or intravenously for 21 days as part of standard of care. Dose, route, and duration determined by treating physician according to clinical condition and guidelines.

SUMMARY:
The CASH study is a randomized, double-blind, placebo-controlled trial evaluating whether adding cilostazol to standard nimodipine therapy improves neurological outcomes in patients with aneurysmal subarachnoid hemorrhage (aSAH). The primary objective is to assess functional outcome at 6 months using the modified Rankin Scale. A total of 630 patients will be enrolled within 96 hours of aSAH onset and treated for 14 days. The study is conducted across 9 centers in France, funded by a PHRC, and overseen by an independent monitoring board.

DETAILED DESCRIPTION:
The CASH trial (Cilostazol in Aneurysmal Subarachnoid Hemorrhage) is a multicenter, randomized, double-blind, placebo-controlled Phase III clinical trial investigating whether the addition of cilostazol to standard nimodipine therapy improves long-term neurological outcomes in patients suffering from aneurysmal subarachnoid hemorrhage (aSAH).

Secondary brain injury following aSAH, particularly delayed cerebral ischemia (DCI) and vasospasm, remains a major cause of mortality and long-term disability. Currently, nimodipine is the only drug with proven efficacy in improving neurological outcomes after aSAH. However, emerging data-mostly from studies conducted in Japan-suggest that cilostazol, a selective phosphodiesterase 3 (PDE3) inhibitor with antiplatelet and vasodilatory effects, may further reduce the risk of ischemic complications and disability when added to standard care.

The cilostazol mechanism includes inhibition of platelet aggregation via cAMP enhancement, vasodilation via nitric oxide release, and endothelial protection. Experimental studies also suggest neuroprotective effects such as attenuation of cortical spreading depolarizations and inhibition of vascular smooth muscle cell proliferation.

The trial will enroll 630 adult patients admitted to intensive care units within 96 hours of a confirmed aSAH due to a ruptured aneurysm that has been secured by either surgical clipping or endovascular coiling. Patients will be randomly assigned to receive either cilostazol 100 mg twice daily for 14 days (administered orally or via gastric tube) or placebo, alongside the standard 21-day nimodipine regimen.

The primary endpoint is the neurological outcome at 6 months, assessed by the modified Rankin Scale (mRS). Secondary outcomes include cognitive performance (MoCA score), return to work, independence in daily activities, hospital and ICU stay durations, 28-day mortality, and incidence of DCI, vasospasm, and cerebral infarctions as defined by imaging or clinical criteria.

The study will be conducted over 49 months (42 months of enrollment + 6 months of follow-up), across 9 French centers, with an expected inclusion rate of 1.9 patients per center per month. Two interim analyses are planned. The study is funded by a Programme Hospitalier de Recherche Clinique (PHRC) and monitored by an independent data safety monitoring board (DSMB).

While cilostazol is generally well tolerated, especially in short-term use, potential side effects include headache, palpitations, diarrhea, arrhythmias, bleeding, and allergic reactions. Previous short-term studies suggest an acceptable safety profile in aSAH patients.

If positive, the CASH study may significantly impact clinical guidelines by supporting the inclusion of cilostazol as an adjunct therapy in the management of aneurysmal subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to an ICU with SAH related to a ruptured cerebral aneurysm occurring within the last 96 hours.
* Aneurysm successfully secured by surgical clipping or endovascular coiling
* Consent of the patient or, if not possible, from a proxy (emergency clause).
* Registration in a national health care system

Exclusion Criteria:

* - Precritical modified Rankin Scale (mRS) > 2
* Nonaneurysmal SAH
* Delayed >96h admission after first symptoms of SAH
* Coma defined by GCS of 3-5 with untreatable aneurysm will be excluded"
* Known allergy to cilostazol
* Pregnancy
* Pre-existing major hepatic, renal, pulmonary or cardiac disease
* Concomitant use of one other anti-platelet and/or anticoagulant agent
* SAH diagnosed on Lumbar puncture with no evidence of blood on CT.
* Tutelage or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-12-14 (Estimated); Study Completion 2029-12-14 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) Score at 6 Months After Aneurysmal Subarachnoid Hemorrhage | At 6 months after aneurysmal subarachnoid hemorrhage
  Neurological functional outcome will be measured using the modified Rankin Scale (mRS) at 6 months post-aneurysmal subarachnoid hemorrhage.
  The mRS is a 7-point ordinal scale ranging from 0 (no symptoms) to 6 (death), assessing the degree of disability or dependence in daily activities.

SECONDARY OUTCOMES:
Functional Outcome at 6 Months Measured by the Subarachnoid Hemorrhage Outcome Tool (SAHOT) | 6 months
  SAHOT total score (range: 0-100; higher scores indicate better functional outcome).
In-hospital morbidity and mortality | 28 days
  Length of stay in Intensive Care Unit (ICU) Length of hospital stay 28-day mortality
Clinical and radiological events predictive of functional status | 6 months
  Delayed cerebral ischemia (DCI): focal neurological deficit or a decrease of at least 2 points in the Glasgow Coma Scale, not occurring immediately after aneurysm occlusion and not attributable to other causes.
  Cerebral vasospasm: reduction in the calibre of proximal cerebral vessels seen on CT angiography, MR angiography, or catheter angiography (DSA), classified according to severity.
  Cerebral infarcts: diagnosis by CT or MRI scan within 6 weeks (or latest imaging before death within 6 weeks, or at autopsy), not present on the CT or MRI scan performed between 24 and 48 hours after early aneurysm occlusion and not attributable to other causes.
Incidence of Cilostazol-Related Major and Minor Adverse Events | 6 months.
  Major adverse events: arrhythmia, abnormal bleeding, allergy.
  Minor adverse events: tachycardia, fever, fainting, nausea, vomiting, stomach pain.
  Notes: Data will be collected from patient reports, clinical assessments, and medical records to evaluate the safety and tolerability of cilostazol.
Cognitive Function at 6 Months Measured by the Montreal Cognitive Assessment (MoCA) | 6 months
  MoCA total score (range: 0-30; higher scores indicate better cognitive function).
Return to Work at 6 Months | 6 months
  Number of participants who have returned to work (yes/no).
Activities of Daily Living (ADL) at 6 Months | 6 months
  Independence in basic self-care activities (scored as dependent/independent).
Instrumental Activities of Daily Living (IADL) at 6 Months | 6 months
  Independence in instrumental daily activities (scored as dependent/independent).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline SCHIMPF, Doctor, Study Chair — Chef de service Anesthésie - Réanimation GHU Paris - Neuro Sainte-Anne; Aurélien MAZERAUD, DOCTOR, Principal Investigator — Anesthésie - Réanimation GHU Paris - Neuro Sainte-Anne

IPD SHARING:
Plan to Share IPD: No
The data will be used exclusively for the analyses planned in the protocol and will not be shared outside the study investigators.

DOCUMENTS (1):
  • Study Protocol (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT07144956/Prot_000.pdf